CLINICAL TRIAL: NCT02219217
Title: Pharmacokinetics of DOLUTEGRAVIR Once Daily and ELVITEGRAVIR/COBICISTAT Once Daily Over 10 Days Following Drug Intake Cessation in Healthy Volunteers
Brief Title: SSAT061: PK of DTG and EVT/COBI in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SSAT061
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir; elvitegravir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No arms (Experimental): All participants will be administered Tivicay® (dolutegravir 50 mg once daily) for 10 days, then will undergo a nine-day wash out period and then take Stribild® (245 mg of tenofovir disoproxil, 200 mg of emtricitabine, 150 mg of elvitegravir and 150 mg of cobicistat) for 10 days.
  Interventions: Drug: Dolutegravir, Elvitegravir and Cobicistat

INTERVENTIONS:
Drug: Dolutegravir, Elvitegravir and Cobicistat

SUMMARY:
The purpose of the study is to look at the levels of three HIV medications: dolutegravir, elvitegravir and cobicistat in blood after the drug intake has been stopped in order to understand how long these drugs persist in the blood. The study will specifically look at blood levels of these three drugs after taking them every day for 10 days dolutegravir on a first stage and a combination of elitegravir and cobicistat in a second stage.

If the participant decides to take part, the duration of the study will be up to 38 days plus a screening visit which will take place up to 28 days prior to the start of the study, and a follow up visit which takes place 7 to 14 days after the last dose of study medication.

This study is not randomised which means that all participants will receive all study medications in the same order. The participant and the study doctor will know which study medications the participant is taking at all times during the study.

ELIGIBILITY:
Inclusion Criteria

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
* Male or non-pregnant, non-lactating females
* Between 18 to 65 years, inclusive
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
* ALT, alkaline phosphatase and bilirubin 1.5xULN (isolated bilirubin greater 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin lesser than 35 per cent). A single repeat is allowed for eligibility determination.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 12 weeks after the study

A female may be eligible to enter and participate in the study if she:

* is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
* is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy: (please see protocol)
* Willing to consent to their personal details being entered onto the TOPS database
* Willing to provide proof of identity by photographic ID at screen and any subsequent visit
* Registered with a GP in the UK

Exclusion Criteria

* Any clinically significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Positive blood screen for hepatitis B surface antigen or C antibodies
* Positive blood screen for HIV-1 or 2 by antibody/antigen assay
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History or presence of allergy to DTG or excipients (D-Mannitol, Microcystalline Cellulose, Povidone, Croscarmellose Sodium, Sodium Stearyl Fumarate, Talc, white film coat)
* Current or recent (within 3 months) gastrointestinal disease
* Known intolerance of lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
* Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
* Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within 3 months of first dose of study drug
* Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
* Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of dolutegravir and elvitegravir/cobicistat after drug intake cessation up to 216 hours post-dose. | 216 hours
  On days 10 and 29: Serial blood specimens will be obtained from each participant for determining drug concentrations of dolutegravir or elvitegravir /cobicistat at the following time points: pre dose (within 10 minutes before dosing), 2, 4, 8 and 12 hours post dose (+/- 5 minutes time window for all post dose time points).
  On days 11-12 and 30-31: Participants will have to attend the unit twice each day, in the mornings and evenings to provide the 24, 36, 48 and 60 hour post dose samples respectively, in order to determine drug concentrations.
  On days 13 to 19 and 32 to 38: Blood will be drawn at the following time points: 72, 96, 120, 144, 168, 192 and 216 hours post last drug dose (dolutegravir and elvitegravir/cobicistat respectively).

CONTACTS AND LOCATIONS:
Locations (1):
- St Stephen's AIDS Trust, London, London, United Kingdom